CLINICAL TRIAL: NCT00002237
Title: Phase I Placebo-Controlled Study of Oral BCX-34 (Peldesine) in HIV-Infected Patients
Brief Title: A Study of Peldesine (BCX-34) in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 301A; 96-009
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-09

CONDITIONS: HIV Infections
Keywords: Placebos; Administration, Oral; Anti-HIV Agents; Viral Load; peldesine
MeSH Terms: conditions — HIV Infections | interventions — peldesine

INTERVENTIONS:
Drug: Peldesine

SUMMARY:
The purpose of this study is to determine the highest amount of peldesine that is safe. This study will also see if this amount of peldesine is effective in lowering HIV levels in the blood.

DETAILED DESCRIPTION:
Patients are given either BCX-35 or placebo for 14 or 28 days. Plasma viral load will be determined at the MTD.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 cell count greater than or equal to 300 cells/mm3 on 3 occasions prior to protocol treatment.
* Plasma viral load by Roche Amplicor HIV Monitor assay greater than or equal to 2,000 RNA copies/ml and less than or equal to 50,000 RNA copies/ml on at least 2 occasions prior to protocol treatment.
* Normal or non-diagnostic electrocardiogram.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Severe opportunistic infection or any other medical condition which in the opinion of the investigators is a contraindication to enrolling in this trial.
* Severe lactose intolerance.

Concurrent Medication:

Excluded:

Concomitant therapy with other medications having primary renal excretion (other than 3TC, ddC, and d4T).

Prior Medication:

Excluded:

* Ongoing dideoxyinosine or other antiretroviral therapy except ZDV, 3TC, ddC, d4T, saquinavir, ritonavir, indinavir, and nelfinavir within 2 weeks of study.
* Participation in a study of any systemic experimental drug within the last 2 months.

Required:

- Ongoing (at least 4 weeks) stable dosage of zidovudine (ZDV) and lamivudine (3TC), ZDV and stavudine (d4T), ZDV and zalcitabine (ddC), d4T and 3TC, ZDV alone, or ddC alone, or in combination with saquinavir, ritonavir, indinavir, or nelfinavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Francis Mem Hosp / HIV Care Unit, San Francisco, California, United States

REFERENCES:
- [Derived] Mboup A, Diabate S, Behanzin L, Guedou FA, Zannou DM, Keke RK, Bachabi M, Gangbo F, Marzinke MA, Hendrix C, Gagnon MP, Alary M. Determinants of HIV Preexposure Prophylaxis Adherence Among Female Sex Workers in a Demonstration Study in Cotonou, Benin: A Study of Behavioral and Demographic Factors. Sex Transm Dis. 2021 Aug 1;48(8):565-571. doi: 10.1097/OLQ.0000000000001373. PMID 33448731
- [Derived] Mboup A, Behanzin L, Guedou FA, Geraldo N, Goma-Matsetse E, Giguere K, Aza-Gnandji M, Kessou L, Diallo M, Keke RK, Bachabi M, Dramane K, Geidelberg L, Cianci F, Lafrance C, Affolabi D, Diabate S, Gagnon MP, Zannou DM, Gangbo F, Boily MC, Vickerman P, Alary M. Early antiretroviral therapy and daily pre-exposure prophylaxis for HIV prevention among female sex workers in Cotonou, Benin: a prospective observational demonstration study. J Int AIDS Soc. 2018 Nov;21(11):e25208. doi: 10.1002/jia2.25208. PMID 31291057